CLINICAL TRIAL: NCT05605912
Title: Efficacy of the Myosuit for Increasing Daily Life Gait Performance in the Home and Community Setting and Gait Capacity in People With Incomplete Spinal Cord Injury
Brief Title: Myosuit in Incomplete Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sint Maartenskliniek (Other)
Responsible Party: Principal Investigator, Noel Keijsers, Prof N.L.W Keijsers, Sint Maartenskliniek
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1033; NL80641.091.22 (Other: CCMO)
Record Dates: First submitted 2022-10-19; First posted 2022-11-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Incomplete Spinal Cord Injury
Keywords: Myosuit; Exosuit; Rehabilitation; Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myosuit intervention (Experimental): Participants perform Myosuit training sessions. After the clinical Myosuit training program, participants receive the Myosuit at their disposal at home for six weeks and a recommendation for physical activity at home.
  Interventions: Device: Myosuit
- Control (Active Comparator): Participants perform conventional training sessions. After the clinical training program, participants receive a recommendation for physical activity at home. After the conventional training program the control group will receive the Myosuit intervention.
  Interventions: Other: Control; Device: Myosuit

INTERVENTIONS:
Other: Control — Participants perform five one-hour conventional training sessions at the Sint Maartenskliniek in which they perform functional exercises. After the conventional training program, the control group will receive a recommendation for physical activity at home for six weeks.
  Arms: Control
Device: Myosuit — Participants perform five one-hour Myosuit training sessions at the Sint Maartenskliniek in which they perform functional exercises and learn to don, doff and use the device for standing, walking, climbing the stairs and sit-to-stand transitions. After the clinical Myosuit training program, participants receive the Myosuit at their disposal at home and a recommendation for physical activity at home for six weeks.
  Other Names: Myoswiss

SUMMARY:
The Myosuit is a light-weighted lower extremity soft exosuit which provide assistance during walking. In this study the Myosuit will be tested in the home and community setting in patients with incomplete spinal cord injury.

DETAILED DESCRIPTION:
Rationale: People with incomplete spinal cord injury (iSCI) show often impairments and limitations related to gait, which negatively affects daily life gait performance (i.e. ambulation in home and community setting) and quality of life. As a consequence of limited gait capacity, these people are likely to develop a sedentary lifestyle resulting in a vicious circle, causing a further decline in gait capacity and daily life gait performance. One of the potential options to improve gait is the use of assistive technology, such as exoskeletons or exosuits. People with iSCI have voluntary control of the leg muscles may benefit more from light-weighted exosuits which provide assistance during walking. Recently, a lower extremity soft exosuit, the Myosuit (MyoSwiss AG), has been introduced. In a small sample study, participants showed an increased gait speed when using the Myosuit compared to their baseline gait speed. Moreover, only a small number of training sessions was required to use the Myosuit. Hence, the Myosuit seems to have a high potential to increase gait capacity and daily life gait performance in people with residual gait capacity.

Objective: The study consists of two parts, randomized controlled trial (RCT) and experimental design. In the RCT, the primary objective is to test the efficacy of the Myosuit for increasing daily life gait performance in the home and community setting in people with iSCI. Secondary, the efficacy of the Myosuit program on gait capacity and its cost-utility will be investigated. Finally, the usability of the Myosuit for use in home and community setting will be evaluated. In the experimental design, we will investigate differences in gait capacity with and without wearing the Myosuit in people with iSCI, by conducting clinical tests. Secondary, differences in gait capacity measured on an instrumented treadmill with and without wearing the Myosuit will be examined.

Study design: RCT and within subject experiment.

Study population: Thirty-four people with chronic iSCI (>6 months after injury) and reduced gait capacity due to reduced knee and/or hip strength (MRC<5) will be recruited for this study. People with iSCI will be included when having an injury level of C or D on the American Spinal Injury Association Impairment Scale. In addition, participants need to have sufficient hand function to don and doff the Myosuit or they need a caregiver who is available to help the participant to use the Myosuit at home. Patients who have another (neurological) disease which can influence motor performance and/or patients who have small wounds, which can be worsened by wearing the Myosuit will be excluded. For the second objective of the experimental design, only people who are be able to walk consecutively for two minutes on a treadmill without any assistive device and without using the handrails will be included.

Intervention: RCT: The intervention group will perform training sessions with the Myosuit at the Sint Maartenskliniek. Thereafter, they will receive the Myosuit at their disposal at home and a recommendation for physical activity for six weeks. The control group will receive a program of conventional physiotherapy at the Sint Maartenskliniek. Thereafter, they receive a recommendation for physical activity for at home for six weeks.

Experimental design: Participants perform clinical tests and measurements on an instrumented treadmill with and without the Myosuit.

Measurements intervention and control group:

* Baseline: Week 1 (T0)
* After clinical training program at the Sint Maartenskliniek: Week 5 (T1)
* During 6 weeks home period: Week 6, 8, 11 (T2, T3, T4)
* After the 6 weeks home period: Week 12 (T5)

Additional measurements for the control group who receive the Myosuit intervention after the conventional program:

* After clinical training program at the Sint Maartenskliniek: Week 16 (T6)
* During 6 weeks home period: Week 17, 19, 22 (T7, T8, T9)
* After the 6 weeks home period: Week 23 (T10)

ELIGIBILITY:
Inclusion Criteria:

* People with a stable chronic iSCI (>6 months after injury).
* Having an injury level of C or D on the American Spinal Injury Association Impairment Scale.
* Age ≥ 18 years.
* Need to have sufficient hand function and standing balance to don and doff the Myosuit or they need a caregiver who is available to help the participant to use the Myosuit at home.
* Having reduced gait capacity due to reduced knee and/or hip strength (MRC=<4).
* Must be able to stand up from a chair without deviating to the left or right side for more than 45 degrees during the movement.
* Can walk for 10 meter without the assistance of another person but can be assisted by assistive devices except knee orthoses.
* People aim to improve walking distance, walking speed or gait capacity.
* Sufficient postural control to walk independently (i.e. without assistance of a person, assistive devices are allowed).
* For the second objective of part B of this study, only people who are be able to walk consecutively for two minutes on a treadmill without any assistive device and without using the handrails will be included

Exclusion Criteria:

* Have another (neurological) disease which can influence motor performance.
* Have wounds which can be worsened by wearing the Myosuit will be excluded.
* Taller than 195 and smaller than 150 cm.
* Body weight of more than 110 kg or less than 45 kg.
* Pregnancy.
* Insufficient mastery of the Dutch language
* Psychiatric background.
* Flexion contracture in knee or hip in excess of 10 degrees.
* Knee varus malposition in excess of 10 degrees or knee valgus malposition in excess of 10 degrees.
* Oncological spinal cord injury.
* Unsuitable for participation according to the rehabilitation physician or researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline daily life gait performance to the home period as assessed by walking time per day (minutes) | Baseline: Week 1 (T0), During the 6-week home period: average over week 6, 8, 11 (T2, T3, T4)
  Measured by the Activ8 for 7 days. At baseline (T0) 7 days are averaged to calculate mean walking time per day. During the 6-week home period all days are averaged to calculate mean walking time per day. (RCT)
Change in preferred walking speed between with and without Myosuit as assessed by the 10 meter walk test (m/s) | After the clinical training program: Week 5 (Myosuit intervention, T1) or week 16 (Control, T6)
  Measure for gait capacity. (experimental design)

SECONDARY OUTCOMES:
Daily life gait performance as assessed by gait quality | Baseline: Week 1 (T0), During the 6-week home period: week 6 and 11 (T2, T4) and week 17 and 22 (T7, T9)
  Measured by inertial measurement units. (RCT)
Change from baseline preferred walking speed at T5 as assessed by the 10 meter walk test (m/s) | Baseline: Week 1 (T0), After the 6-week home period: Week 12 and 23 (T5, T10)
  Measure for gait capacity. (RCT)
Maximum walking speed as assessed by the 10 meter walk test (m/s) | Baseline: Week 1 (T0), After the 6-week home period: Week 12 and 23 (T5, T10)
  Measure for gait capacity. (RCT)
Walking speed as assessed by the 6 minutes walk test (m/s) | Baseline: Week 1 (T0), After the 6-week home period: Week 12 and 23 (T5, T10)
  Measure for gait capacity. (RCT)
Functional ambulation as assessed by the spinal cord injury functional ambulation profile (SCI-FAP) | Baseline: Week 1 (T0), After the 6-week home period: Week 12 and 23 (T5, T10)
  Measure for gait capacity. The SCI-FAP is composed of 7 tasks: carpet, up & go, obstacles, stairs, carry, step, and door. The highest total score is 2100. The SCI-FAP is a timed measure, a low score indicates better function. (RCT)
Usability as assessed by the System Usability Scale (SUS) | After the clinical training program: Week 5 and 16 (T1, T6), After the 6-week home period: Week 12 and 23 (T5, T10)
  The range is between 0 and 100, with a higher score indicating better usability. (RCT)
Usability as assessed by the Dutch version of the quebec user evaluation of satisfaction with assistive technology (D-QUEST) | After the clinical training program: Week 5 and 16 (T1, T6), After the 6-week home period: Week 12 and 23 (T5, T10)
  The range is between 1 and 5, with a higher score indicating greater satisfaction. (RCT)
Quality-adjusted-life years gain assessed by EuroQol five-dimension scale questionnaire (EQ5D-5L) | Baseline: Week 1 (T0), After the 6-week home period: Week 12 and 23 (T5, T10)
  Measure for quality of life to investigate cost-utility. The EQ5D-5L consists of five levels with a maximum score of 1 which indicates the best health state. In addition there is a visual analogue scale with a maximum score of 100 to indicate general health status. (RCT)
General and Disease Specific Self-efficacy Scale | Baseline: Week 1 (T0), After the 6-week home period: Week 12 and 23 (T5, T10)
  Questionnaire contains confidence in general, confidence in managing with your physical condition and confidence in walking. The range is between 0 and 160, with a higher score indicating higher confidence. (RCT)
Maximum walking speed as assessed by the 10 meter walk test (m/s) | After the clinical training program: Week 5 and 16 (T1, T6)
  Measure for gait capacity. (experimental design)
Walking speed as assessed by the 6 minutes walk test (m/s) | After the clinical training program: Week 5 and 16 (T1, T6)
  Measure for gait capacity. (experimental design)
Preferred walking speed as assessed by walking on the GRAIL (m/s) | After the clinical training program: Week 5 and 16 (T1, T6)
  Measure for gait capacity. Preferred walking speed is measured during 2 minutes self-paced walking on the GRAIL. (experimental design)
Step length as assessed by walking on the GRAIL | After the clinical training program: Week 5 and 16 (T1, T6)
  Measure for gait capacity. Step length is measured during 2 minutes walking on fixed speed on the GRAIL. (experimental design)
Step time as assessed by walking on the GRAIL | After the clinical training program: Week 5 and 16 (T1, T6)
  Measure for gait capacity. Step time is measured during 2 minutes walking on fixed speed on the GRAIL. (experimental design)
Ankle range of motion as assessed by walking on the GRAIL | After the clinical training program: Week 5 and 16 (T1, T6)
  Measure for gait capacity. Ankle range of motion is measured during 2 minutes walking on fixed speed on the GRAIL. (experimental design)
Maximum ankle plantar flexion as assessed by walking on the GRAIL | After the clinical training program: Week 5 and 16 (T1, T6)
  Measure for gait capacity. Maximum ankle plantar flexion is measured during 2 minutes walking on fixed speed on the GRAIL. (experimental design)
Knee range of motion as assessed by walking on the GRAIL | After the clinical training program: Week 5 and 16 (T1, T6)
  Measure for gait capacity. Knee range of motion is measured during 2 minutes walking on fixed speed on the GRAIL. (experimental design)
Maximum knee extension as assessed by walking on the GRAIL | After the clinical training program: Week 5 and 16 (T1, T6)
  Measure for gait capacity. Maximum knee extension is measured during 2 minutes walking on fixed speed on the GRAIL. (experimental design)
Hip range of motion as assessed by walking on the GRAIL | After the clinical training program: Week 5 and 16 (T1, T6)
  Measure for gait capacity. Hip range of motion is measured during 2 minutes walking on fixed speed on the GRAIL. (experimental design)
Maximum hip extension as assessed by walking on the GRAIL | After the clinical training program: Week 5 and 16 (T1, T6)
  Measure for gait capacity. Maximum hip extension is measured during 2 minutes walking on fixed speed on the GRAIL. (experimental design)
Variable error of the precision stepping task as assessed by walking on the GRAIL | After the clinical training program: Week 5 and 16 (T1, T6)
  Measure for gait adaptability. (experimental design)

OTHER OUTCOMES:
Sex (man/woman) | Baseline: Week 1 (T0)
  Descriptive outcome measure.
Age (years) | Baseline: Week 1 (T0)
  Descriptive outcome measure.
Height (cm) | Baseline: Week 1 (T0)
  Descriptive outcome measure.
Weight (kg) | Baseline: Week 1 (T0)
  Descriptive outcome measure.
Body Mass Index | Baseline: Week 1 (T0)
  Descriptive outcome measure. Calculated with weight and height.
Time since spinal cord injury (years) | Baseline: Week 1 (T0)
  Descriptive outcome measure.
Spinal cord injury classification defined by the American Spinal Injury Association (ASIA) impairment scale (C or D) | Baseline: Week 1 (T0)
  Descriptive outcome measure. The scale has five classification levels (A-E), ranging from complete loss of neural function (A) in the affected area to completely normal (E).
Level of spinal cord injury | Baseline: Week 1 (T0)
  Descriptive outcome measure. There are four sections that impact the level of spinal cord injury: cervical, thoracic, lumbar and sacral.
Muscle strength as assessed by Medical Research Council (MRC) scale | Baseline: Week 1 (T0)
  Descriptive outcome measure. Range from 0 - 5 with higher scores indicating more strength
Spasticity as assessed by Modified Ashworth Scale (MAS) | Baseline: Week 1 (T0)
  Descriptive outcome measure. Range from 0 - 4 with higher scores indicating more spasticity
Sensory function as assessed by the American Spinal Cord Injury Association (ASIA) Impairment Scale | Baseline: Week 1 (T0)
  Descriptive outcome measure. Range from 0 - 2 with lower scores indicating more impaired sensory function

CONTACTS AND LOCATIONS:
Overall Officials: Bart van den Bemt, Principal Investigator — Sint Maartenskliniek
Locations (1):
- Sint Maartenskliniek, Ubbergen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balasubramanian CK, Clark DJ, Fox EJ. Walking adaptability after a stroke and its assessment in clinical settings. Stroke Res Treat. 2014;2014:591013. doi: 10.1155/2014/591013. Epub 2014 Aug 28. PMID 25254140
- [Background] DiPiro ND, Holthaus KD, Morgan PJ, Embry AE, Perry LA, Bowden MG, Gregory CM. Lower Extremity Strength Is Correlated with Walking Function After Incomplete SCI. Top Spinal Cord Inj Rehabil. 2015 Spring;21(2):133-9. doi: 10.1310/sci2102-133. Epub 2015 Apr 12. PMID 26364282
- [Background] Fanchamps MHJ, Horemans HLD, Ribbers GM, Stam HJ, Bussmann JBJ. The Accuracy of the Detection of Body Postures and Movements Using a Physical Activity Monitor in People after a Stroke. Sensors (Basel). 2018 Jul 5;18(7):2167. doi: 10.3390/s18072167. PMID 29976900
- [Background] Haufe FL, Kober AM, Schmidt K, Sancho-Puchades A, Duarte JE, Wolf P, Riener R. User-driven walking assistance: first experimental results using the MyoSuit. IEEE Int Conf Rehabil Robot. 2019 Jun;2019:944-949. doi: 10.1109/ICORR.2019.8779375. PMID 31374751
- [Background] Haufe FL, Schmidt K, Duarte JE, Wolf P, Riener R, Xiloyannis M. Activity-based training with the Myosuit: a safety and feasibility study across diverse gait disorders. J Neuroeng Rehabil. 2020 Oct 8;17(1):135. doi: 10.1186/s12984-020-00765-4. PMID 33032627
- [Background] Horemans H, Kooijmans H, van den Berg-Emons R, Bussmann H. The Activ8 activity monitor: Validation of posture and movement classification. J Rehabil Assist Technol Eng. 2020 Mar 16;7:2055668319890535. doi: 10.1177/2055668319890535. eCollection 2020 Jan-Dec. PMID 32206335
- [Background] Ishikawa S, Stevens SL, Kang M, Morgan DW. Reliability of daily step activity monitoring in adults with incomplete spinal cord injury. J Rehabil Res Dev. 2011;48(10):1187-94. doi: 10.1682/jrrd.2010.09.0190. PMID 22234663
- [Background] Just IA, Fries D, Loewe S, Falk V, Cesarovic N, Edelmann F, Feuerstein A, Haufe FL, Xiloyannis M, Riener R, Schoenrath F. Movement therapy in advanced heart failure assisted by a lightweight wearable robot: a feasibility pilot study. ESC Heart Fail. 2022 Jun;9(3):1643-1650. doi: 10.1002/ehf2.13903. Epub 2022 Mar 23. PMID 35320878
- [Background] Lankhorst K, van den Berg-Emons RJ, Bussmann JBJ, Horemans HLD, de Groot JF. A Novel Tool for Quantifying and Promoting Physical Activity in Youths With Typical Development and Youths Who Are Ambulatory and Have Motor Disability. Phys Ther. 2019 Mar 1;99(3):354-363. doi: 10.1093/ptj/pzy152. PMID 30649497
- [Background] Maetzler W, Rochester L, Bhidayasiri R, Espay AJ, Sanchez-Ferro A, van Uem JMT. Modernizing Daily Function Assessment in Parkinson's Disease Using Capacity, Perception, and Performance Measures. Mov Disord. 2021 Jan;36(1):76-82. doi: 10.1002/mds.28377. Epub 2020 Nov 15. PMID 33191498
- [Background] Muthukrishnan N, Abbas JJ, Krishnamurthi N. A Wearable Sensor System to Measure Step-Based Gait Parameters for Parkinson's Disease Rehabilitation. Sensors (Basel). 2020 Nov 10;20(22):6417. doi: 10.3390/s20226417. PMID 33182658
- [Background] Mohamed Refai MI, van Beijnum BF, Buurke JH, Veltink PH. Portable Gait Lab: Tracking Relative Distances of Feet and CoM Using Three IMUs. IEEE Trans Neural Syst Rehabil Eng. 2020 Oct;28(10):2255-2264. doi: 10.1109/TNSRE.2020.3018158. Epub 2020 Aug 20. PMID 32816676
- [Background] Saraf P, Rafferty MR, Moore JL, Kahn JH, Hendron K, Leech K, Hornby TG. Daily stepping in individuals with motor incomplete spinal cord injury. Phys Ther. 2010 Feb;90(2):224-35. doi: 10.2522/ptj.20090064. Epub 2009 Dec 18. PMID 20022997
- [Background] Schmidt K, Duarte JE, Grimmer M, Sancho-Puchades A, Wei H, Easthope CS, Riener R. The Myosuit: Bi-articular Anti-gravity Exosuit That Reduces Hip Extensor Activity in Sitting Transfers. Front Neurorobot. 2017 Oct 27;11:57. doi: 10.3389/fnbot.2017.00057. eCollection 2017. PMID 29163120
- [Background] Ummels D, Beekman E, Theunissen K, Braun S, Beurskens AJ. Counting Steps in Activities of Daily Living in People With a Chronic Disease Using Nine Commercially Available Fitness Trackers: Cross-Sectional Validity Study. JMIR Mhealth Uhealth. 2018 Apr 2;6(4):e70. doi: 10.2196/mhealth.8524. PMID 29610110
- [Background] van der Salm A, Nene AV, Maxwell DJ, Veltink PH, Hermens HJ, IJzerman MJ. Gait impairments in a group of patients with incomplete spinal cord injury and their relevance regarding therapeutic approaches using functional electrical stimulation. Artif Organs. 2005 Jan;29(1):8-14. doi: 10.1111/j.1525-1594.2004.29004.x. PMID 15644078
- [Background] van Dijsseldonk RB, de Jong LAF, Groen BE, Vos-van der Hulst M, Geurts ACH, Keijsers NLW. Gait Stability Training in a Virtual Environment Improves Gait and Dynamic Balance Capacity in Incomplete Spinal Cord Injury Patients. Front Neurol. 2018 Nov 20;9:963. doi: 10.3389/fneur.2018.00963. eCollection 2018. PMID 30524356
- [Background] van Uem JM, Marinus J, Canning C, van Lummel R, Dodel R, Liepelt-Scarfone I, Berg D, Morris ME, Maetzler W. Health-Related Quality of Life in patients with Parkinson's disease--A systematic review based on the ICF model. Neurosci Biobehav Rev. 2016 Feb;61:26-34. doi: 10.1016/j.neubiorev.2015.11.014. Epub 2015 Dec 2. PMID 26645499
- [Derived] Visch L, Groen BE, Geurts ACH, van Nes IJW, Keijsers NLW. Effect of a soft exosuit on daily life gait performance in people with incomplete spinal cord injury: study protocol for a randomized controlled trial. Trials. 2024 Sep 6;25(1):592. doi: 10.1186/s13063-024-08412-2. PMID 39242508
- See also: Link to the research project website — https://www.maartenskliniek.nl/research-innovation-en/research-innovation-projects/efficacy-of-the-myosuit